CLINICAL TRIAL: NCT00235534
Title: Immediate Versus Delayed Initiation of Oral Contraceptive Pills After Therapeutic Abortion - A Randomized Trial
Brief Title: Trial of Immediate Versus Delayed Initiation of Oral Contraceptive Pills After Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H11779-26464-01
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Abortion
Keywords: abortion; randomized; contraception; pregnancy; compliance; continuation; oral contraceptive pills
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Immediate start (Experimental): Initiate selected birth control method before leaving the clinic at the time of the abortion procedure.
  Interventions: Behavioral: Immediate initiation of OCPs
- Sunday start (Active Comparator): Begin birth control the first Sunday after leaving the clinic
  Interventions: Behavioral: Delayed initiation of OCPs

INTERVENTIONS:
Behavioral: Immediate initiation of OCPs
  Arms: Immediate start
Behavioral: Delayed initiation of OCPs
  Arms: Sunday start

SUMMARY:
This is a randomized, controlled trial investigating whether immediate versus standard, "Sunday Start", initiation of oral contraceptive pills (OCPs) in post-abortion subjects can improve compliance and the continuation of contraception. Immediate initiation of OCPs has been studied in women seeking contraception when they are not immediately post-abortion, and this "Quick Start" method has been shown to improve the continuation of OCPs into a second pill pack. The primary hypothesis of this study is that immediate initiation of OCPs in post-abortal women will improve the continuation of contraception over delayed initiation on the first Sunday after an abortion.

DETAILED DESCRIPTION:
The United States has a higher rate of unintended pregnancy than Canada or any other developed nation in Europe. OCPs are the most common method of hormonal contraception used in this country. Perfect use can lead to failure rates as low as 0.1% per year. Actual failure rates are much higher, often due to non-compliance with OCP use. Several recent studies have examined the "Quick Start", or initiation of OCPs in front of the provider while still at the clinic, regardless of time in the cycle. These studies have shown that women who swallowed the first OCP in the clinic were more likely to continue the OCP into the second month. Women who are seen in clinics for a therapeutic abortion (TAB) are often at extremely high risk for another unintended/unwanted pregnancy. If compliance in OCP use could be improved in this group of women, unintended/unwanted pregnancy rates could be reduced. One concern about the "Quick Start" technique is that women may have already ovulated or conceived when OCPs are initiated mid-cycle. In the post-abortal setting, this is not a concern. Applying the "Quick Start" technique to post-abortion patients and having women take the first of their OCPs while still in the clinic after their abortion may improve compliance and continuation of OCP use.

This is a prospective, randomized, controlled trial in post-abortal women, and will last approximately 24 months. All of the study subjects will receive a single pack of combination OCPs and a one-year prescription after their TAB. The women in the immediate start arm will then take their first OCP in the clinic, observed by clinic staff, before leaving. The controls will be instructed to begin the OCPs on the first Sunday following their abortion. All subjects will receive the same medication with the only difference being the timing of initiation of the OCPs. Measurements of continuation will be determined by telephone interviews administered at two and six months after the subjects' abortion.

ELIGIBILITY:
Inclusion Criteria:

* Any woman aged 13-45 who presents to the Women's Options Clinic and desires to use OCPs for post-abortion contraception.

Exclusion Criteria:

* Gestational age above 23 weeks and 1 day.
* Any absolute contraindication for combination OCP use (smoking > 20 cigarettes a day over age 35, history of venous thromboembolic event or pulmonary embolism, history of or current ischemic heart disease, history of stroke, vascular disease, complicated valvular heart disease [pulmonary hypertension, atrial fibrillation, history of subacute bacterial endocarditis], severe hypertension with blood pressure >160/100, migraines with focal neurologic symptoms, current breast cancer, active viral hepatitis, severe cirrhosis, or benign or malignant liver tumors).
* Patients who speak languages other than English or Spanish.
* Patients who do not have a phone or who have a phone where any contact might compromise the confidentiality of their abortions.

Ages: 13 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2005-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Continuation of OCPs after abortion | Two and six months post-enrollment
  Assessed by phone survey

SECONDARY OUTCOMES:
Compliance with OCPs after abortion | Two and six months post-enrollment
  assessed by phone survey
Bleeding patterns on OCPs after abortion | Two months post-abortion
  assessed by phone survey
Satisfaction with OCPs after abortion | six months post-enrollment
  assessed by phone survey

CONTACTS AND LOCATIONS:
Overall Officials: Jody E Steinauer, MD, MAS, Principal Investigator — University of California, San Francisco; Sarah W Prager, MD, Study Director — University of California, San Francisco
Locations (1):
- Women's Options Clinic at San Francisco General Hospital, San Francisco, California, United States